CLINICAL TRIAL: NCT03491319
Title: Cephalic Spread of Block With Head Down Tilt in Spinal Anaesthesia - A Randomised Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nitte University (Other)
Responsible Party: Principal Investigator, Dr. Sara Jaison, Junior Resident, Nitte University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: nitteU
Record Dates: First submitted 2018-03-31; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2017-07

CONDITIONS: Head-Down Tilt Following Spinal Anesthesia
Keywords: Anesthetics, Local; Head-Down Tilt; Anesthesia, Spinal; hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated to one of the 3 groups by closed envelope method
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: First anaesthesiologist performed the spinal anaesthesia, gave table tilt using clinometer according to group allocation and assessed spinal blockade till 10 min after intrathecal injection. Thereafter it was done by the second anaesthesiologist who was blinded to the patient grouping
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C Control (Placebo Comparator): spinal anaesthesia was given with table in neutral positon. Same position was maintained after spinal anaesthesia
  Interventions: Procedure: Group C - neutral
- Group X (Active Comparator): spinal anaesthesia was given with table in neutral positon. 10 degree head low position was maintained for 10 minutes following spinal
  Interventions: Procedure: Group X - head low tilt
- Group Y (Active Comparator): the table was put in 10 degree head low position before proceeding to give spinal anaesthesia. Head low position was maintained for 10 minutes following spinal
  Interventions: Procedure: Group Y - head low tilt

INTERVENTIONS:
Procedure: Group X - head low tilt — spinal anaesthesia was given with table in neutral positon. 10 degree head low position was maintained for 10 minutes following spinal anaesthesia
  Arms: Group X
Procedure: Group Y - head low tilt — the table was put in 10 degree head low position before proceeding to give spinal anaesthesia. Head low position was maintained for 10 minutes following spinal
  Arms: Group Y
Procedure: Group C - neutral — spinal anaesthesia was given with table in neutral positon. Patient was maintained in supine position for 10 minutes following spinal anaesthesia
  Arms: Group C Control

SUMMARY:
Subarachnoid block has become an established and reliable method of providing anaesthesia for lower abdominal and lower limb surgeries. Several factors determine the spread of local anaesthetic solutions in CSF. Among them, patient position is an important determining factor. Anesthesiologists give various degrees of head down tilt which they believe is both safe for the patient and will result in adequate level of block. Often these are arbitrarily done by the operator as most of the operation theatre tables are not equipped with any device to measure the accurate degree of tilt. As there is no agreement on the effect of Trendelenberg position on height of subarachnoid block, the current clinical study will be undertaken to estimate the effect of operation theatre table tilt at the time of lumbar puncture on the height of subarachnoid block.

DETAILED DESCRIPTION:
Subarachnoid block has become an established and reliable method of providing anaesthesia for lower abdominal and lower limb surgeries. A definitive advantage that subarachnoid block provides is the profound nerve block that can be produced in a large part of the body by the relatively simple injection of a small amount of local anaesthetic. Twenty-five factors have been invoked as determinants of the spread of local anaesthetic solutions in CSF. Among them, patient position is an important determining factor.

Operation theatre table tilts have been used to influence the spread of hyperbaric solution to ultimately influence the final height of the block. Studies have shown that a 10 degree head down tilt can result in cephalad spread of analgesia when compared to the horizontal group. So, in cases where the spinal block level was not high enough to perform a given surgery, the Trendelenburg position has been used to extend the level of the block. Hence, it is assumed that a higher level of block can be achieved with a smaller volume of the local anaesthetic agent, thus reducing the side effects. But others have noted that there was no statistically significant increase in the level of block even with 15 degree head down tilt.

In spite of this, anesthesiologists give various degrees of head down tilt which they believe is both safe for the patient and will result in adequate level of block. Often these are arbitrarily done by the operator as most of the operation theatre tables are not equipped with any device to measure the accurate degree of tilt.

An application called clinometer that utilizes the gyroscope sensor and determines the plane of the gadget in vertical as well as horizontal directions has been described. This application can be used to measure the exact degree of tilt given after sub arachnoid block.

As there is no agreement on the effect of Trendelenberg position on height of subarachnoid block, the current clinical study will be undertaken to estimate the effect of operation theatre table tilt at the time of lumbar puncture on the height of subarachnoid block.

ELIGIBILITY:
Inclusion Criteria:

* Patients belonging to ASA physical status I and II undergoing lower abdominal and lower limb surgeries under spinal anaesthesia

Exclusion Criteria:

* Patient refusal
* contraindicated for spinal anaesthesia
* allergy to local anaesthetic agents used
* obesity (body mass index >29 kg/m2)
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Maximum height of block | from 5 minutes to 150 minutes after intrathecal injection
Two segment regression time | from 5 minutes to 150 minutes after intrathecal injection
  time from injection of spinal drug to regression of the sensory block by two segments from the maximum

SECONDARY OUTCOMES:
Hypotension | every minute for 5 min after intrathecal drug administration, every 5 min till 30 min and thereafter every 10 minutes till 150 minutes after intrathecal injection
  drop in systolic blood pressure to less than 30% of baseline values or systolic blood pressure (SBP) below 90mmHg
Tachycardia | every minute for 5 min after intrathecal drug administration, every 5 min till 30 min and thereafter every 10 minutes till 150 minutes after intrathecal injection.
  heart rate more than 100bpm or increase by more than 30% over baseline value.
Bradycardia | every minute for 5 min after intrathecal drug administration, every 5 min till 30 min and thereafter every 10 minutes till 150 minutes after intrathecal injection
  heart rate less than 50bpm or decrease by more than 30% below baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Sripada Mehandale, MBBS, MD, Study Director — Associate Professor

REFERENCES:
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Sinclair CJ, Scott DB, Edstrom HH. Effect of the trendelenberg position on spinal anaesthesia with hyperbaric bupivacaine. Br J Anaesth. 1982 May;54(5):497-500. doi: 10.1093/bja/54.5.497. PMID 7073918
- [Background] Dixit RB, Neema MM. Use of an Android application "clinometer" for measurement of head down tilt given during subarachnoid block. Saudi J Anaesth. 2016 Jan-Mar;10(1):29-32. doi: 10.4103/1658-354X.169471. PMID 26955307
- [Background] Kim JT, Shim JK, Kim SH, Jung CW, Bahk JH. Trendelenburg position with hip flexion as a rescue strategy to increase spinal anaesthetic level after spinal block. Br J Anaesth. 2007 Mar;98(3):396-400. doi: 10.1093/bja/ael370. Epub 2007 Feb 5. PMID 17283005
- [Result] Hocking G, Wildsmith JA. Intrathecal drug spread. Br J Anaesth. 2004 Oct;93(4):568-78. doi: 10.1093/bja/aeh204. Epub 2004 Jun 25. No abstract available. PMID 15220175
- [Result] Miyabe M, Namiki A. The effect of head-down tilt on arterial blood pressure after spinal anesthesia. Anesth Analg. 1993 Mar;76(3):549-52. doi: 10.1213/00000539-199303000-00017. PMID 8452265